CLINICAL TRIAL: NCT07222189
Title: A Multinational, Multicenter Extension Study to Investigate the Long-term Safety, Tolerability and Efficacy of Balinatunfib in Adults With Crohn's Disease or Ulcerative Colitis
Brief Title: A Study to Investigate the Long-term Safety, Tolerability and Efficacy of Balinatunfib in Participants With Crohn's Disease or Ulcerative Colitis (SPECIFI-IBD-LTS)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LTS19689; 2025-522511-42 (Registry Identifier: CTIS); U1111-1321-1765 (Registry Identifier: WHO ICTRP)
Record Dates: First submitted 2025-10-27; First posted 2025-10-29 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Colitis Ulcerative; Crohn's Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding is not applicable for open-label arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- CD cohort: balinatunfib dose regimen 1 (Experimental): Participants will receive balinatunfib dose regimen 1
  Interventions: Drug: balinatunfib
- CD cohort: balinatunfib dose regimen 2 (Experimental): Participants will receive balinatunfib dose regimen 2
  Interventions: Drug: balinatunfib
- CD cohort: balinatunfib dose regimen 3 (Experimental): Participants will receive balinatunfib dose regimen 3
  Interventions: Drug: balinatunfib
- CD cohort: Placebo (Placebo Comparator): Participants will receive balinatunfib-matching placebo
  Interventions: Drug: balinatunfib-matching placebo
- UC cohort: balinatunfib dose regimen 1 (Experimental): Participants will receive balinatunfib dose regimen 1
  Interventions: Drug: balinatunfib
- UC cohort: balinatunfib dose regimen 2 (Experimental): Participants will receive balinatunfib dose regimen 2
  Interventions: Drug: balinatunfib
- UC cohort: balinatunfib dose regimen 3 (Experimental): Participants will receive balinatunfib dose regimen 3
  Interventions: Drug: balinatunfib
- UC cohort: Placebo (Placebo Comparator): Participants will receive balinatunfib-matching placebo
  Interventions: Drug: balinatunfib-matching placebo

INTERVENTIONS:
Drug: balinatunfib — Pharmaceutical form:Tablet -Route of administration:Oral
  Other Names: SAR441566
  Arms: CD cohort: balinatunfib dose regimen 1; CD cohort: balinatunfib dose regimen 2; CD cohort: balinatunfib dose regimen 3; UC cohort: balinatunfib dose regimen 1; UC cohort: balinatunfib dose regimen 2; UC cohort: balinatunfib dose regimen 3
Drug: balinatunfib-matching placebo — Pharmaceutical form:Tablet -Route of administration:Oral
  Arms: CD cohort: Placebo; UC cohort: Placebo

SUMMARY:
LTS19689 is a multinational, multicenter extension study to evaluate the long-term safety, tolerability and efficacy of balinatunfib in participants with Crohn's disease (CD) or ulcerative colitis (UC) who completed the 52-week treatment period (on balinatunfib or placebo) in the parent studies, SPECIFI-CD (DRI18212) or SPECIFI-UC (DRI17822), respectively.

* The primary objective of this study is to assess the long-term safety and tolerability of different doses of balinatunfib in participants with CD or UC, as measured by the number and percentage of participants with CD or UC with treatment emergent adverse events (TEAEs), serious adverse events (SAEs) and adverse events of special interest (AESIs) during the study period.
* The study will consist of 2 independent cohorts through the study given the distinct nature of each disease:

  * CD Cohort: comprised of CD participants enrolled from SPECIFI-CD (DRI18212).
  * UC Cohort: comprised of UC participants enrolled from SPECIFI-UC (DRI17822).
* The study will consist of the following study periods for each cohort:

  * A Double-Blind (DB) treatment period of up to 104 weeks for eligible participants from the DB maintenance phases of the respective parent studies.
  * An Open-Label (OL) treatment period of up to 104 weeks for:

    * Eligible participants from either the DB or OL periods of the parent studies,
    * Eligible participants who meet escape criteria at any time during the DB period of the LTS19689.
  * A 2-week follow-up period following the End of Treatment (EOT). The study duration will be up to 107 weeks, with the treatment duration up to 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

* Participants with Crohn's Disease (CD) or ulcerative colitis (UC) who completed treatment at Week 52 of the SPECIFI-CD (DRI18212) or SPECIFI-UC (DRI17822) studies, respectively:

  * Participants with CD

    1. who complete double-blinded treatment at Week 52 of SPECIFI-CD (DRI18212) study;
    2. who complete open label treatment and achieve the appropriate outcomes at Week 52 of SPECIFI-CD (DRI18212) study.

       OR
  * Participants with UC

    1. who complete double-blinded treatment at Week 52 of SPECIFI-UC (DRI17822) study;
    2. who complete open label treatment and achieve the appropriate outcomes at Week 52 of the SPECIFI-UC (DRI17822) study.
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Women participants should not be pregnant or breastfeeding

Exclusion Criteria:

* Participants with CD who develop a new medical condition precluding participation as described in Exclusion criteria of SPECIFI-CD (DRI18212) clinical trial protocol.
* Participants with UC who develop a new medical condition precluding participation as described in Exclusion criteria of SPECIFI-UC (DRI17822) clinical trial protocol.
* Participants who developed a new medical condition or a change in status of an established medical condition which (per Investigator's medical judgment) would adversely affect the participation in this study or would require permanent IMP discontinuation.
* Participants who permanently discontinued IMP during the parent study or temporarily discontinued IMP for more than 14 consecutive calendar days by the time of Day 1 of LTS19689.
* Participants who, during their participation in the parent study, developed an adverse event (AE) or a serious adverse event (SAE) deemed related to balinatunfib, which in the opinion of the Investigator could indicate that continued treatment with balinatunfib may present an unreasonable risk for the participant.
* Participants who in the parent study had documented nonadherence to IMP or to standard therapies for CD or UC, or who used a prohibited medication concomitant with IMP or during a temporary IMP discontinuation period.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 19 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Estimated)
Dates: Start 2026-05-12 (Estimated); Primary Completion 2030-05-10 (Estimated); Study Completion 2030-05-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Crohn's Disease with treatment emergent adverse events (TEAEs), serious adverse events (SAEs) and adverse events of special interest (AESIs) | Up to End of Study (approximately 106 weeks)
Number of participants with ulcerative colitis with treatment emergent adverse events (TEAEs), serious adverse events (SAEs) and adverse events of special interest (AESIs) | Up to End of Study (approximately 106 weeks)

SECONDARY OUTCOMES:
Proportion of participants with Crohn's Disease in endoscopic remission based on simple endoscopic score for Crohn's disease (SES-CD) | Week 52
  Endoscopic remission is defined as SES-CD ≤4 points (SES CD ≤2 points for isolated ileal disease) and a SES-CD decrease ≥2 points with no SES-CD subscore >1 point from baseline. The SES-CD evaluates 4 endoscopic items (ulcer size, ulcerated surface, affected surface, and narrowing, each on a scale from 0 (none) to 3 in 5 segments assessed during ileocolonoscopy (ileum, right colon, transverse colon, sigmoid and left colon, and rectum). The total score is the sum of the 4 endoscopic variable scores and ranges from 0 to 56, where higher scores indicate more severe disease.
Proportion of participants with Crohn's Disease in endoscopic remission based on simple endoscopic score for Crohn's disease (SES-CD) | Week 104
  Endoscopic remission is defined as SES-CD ≤4 points (SES CD ≤2 points for isolated ileal disease) and a SES-CD decrease ≥2 points with no SES-CD subscore >1 point from baseline. The SES-CD evaluates 4 endoscopic items (ulcer size, ulcerated surface, affected surface, and narrowing, each on a scale from 0 (none) to 3 in 5 segments assessed during ileocolonoscopy (ileum, right colon, transverse colon, sigmoid and left colon, and rectum). The total score is the sum of the 4 endoscopic variable scores and ranges from 0 to 56, where higher scores indicate more severe disease.
Proportion of participants with Crohn's Disease in clinical remission based on Crohn's disease activity index (CDAI) | Week 52
  Clinical remission is defined as CDAI <150. The CDAI score is composed of eight items: 3 of them (abdominal pain, stool frequency and general well-being) completed by the participant and the others (use of anti-diarrheal medications, extraintestinal complications, palpable abdominal mass, hematocrit levels, and body weight) assessed and reported by the clinician. The CDAI is derived from summing up the weighted individual scores of eight items. Scores on the CDAI scale range from 0 to 600, with higher scores indicating more severe disease.
Proportion of participants with Crohn's Disease in clinical remission based on Crohn's disease activity index (CDAI) | Week 104
  Clinical remission is defined as CDAI <150. The CDAI score is composed of eight items: 3 of them (abdominal pain, stool frequency and general well-being) completed by the participant and the others (use of anti-diarrheal medications, extraintestinal complications, palpable abdominal mass, hematocrit levels, and body weight) assessed and reported by the clinician. The CDAI is derived from summing up the weighted individual scores of eight items. Scores on the CDAI scale range from 0 to 600, with higher scores indicating more severe disease.
Proportion of participants with ulcerative colitis in clinical remission based on modified Mayo Score (mMS) | Week 52
  Clinical remission by modified Mayo score (mMS) is defined as a mMS score of 0 to 2, including stool frequency (SF) of 0 or 1, rectal bleeding (RB) subscore of 0, and centrally read modified Mayo Endoscopic Subscore [mMES] of 0 or 1 (score of 1 modified to exclude friability).Each component of the mMS (SF, RB, and mMES) is scored from 0 to 3. The total mMS ranges from 0 to 9 with higher scores indicating greater disease severity
Proportion of participants with ulcerative colitis in clinical remission based on modified Mayo Score (mMS) | Week 104
  Clinical remission by modified Mayo score (mMS) is defined as a mMS score of 0 to 2, including stool frequency (SF) of 0 or 1, rectal bleeding (RB) subscore of 0, and centrally read modified Mayo Endoscopic Subscore [mMES] of 0 or 1 (score of 1 modified to exclude friability).Each component of the mMS (SF, RB, and mMES) is scored from 0 to 3. The total mMS ranges from 0 to 9 with higher scores indicating greater disease severity

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org